CLINICAL TRIAL: NCT01691586
Title: Remote Monitoring of Heart Failure Patients With Cardiovascular Implantable Electronic Device: The Patient Perspective
Brief Title: Patient Perspective on Remote Monitoring of Cardiovascular Implantable Electronic Devices
Acronym: REMOTE-CIED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Boston Scientific Corporation (Industry); Tilburg University (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, M. Meine, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCU.DHL.001
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Congestive Heart Failure
Keywords: implantable defibrillators; remote patient monitoring; patient-reported outcomes; cost-effectiveness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote patient management (Experimental): Remote patient management system + yearly in-clinic follow-up
  Interventions: Device: Remote patient monitoring; Other: In-Clinic check-ups
- In-Clinic follow-up (Other): In-clinic follow-up according to standard practice (every 3-6 months)
  Interventions: Other: In-Clinic check-ups

INTERVENTIONS:
Device: Remote patient monitoring — Remote monitoring of ICD and heart failure data
  Other Names: Boston Scientific LATITUDE system
  Arms: Remote patient management
Other: In-Clinic check-ups — Calender-based In-Clinic ICD check-up

SUMMARY:
A relatively new and promising development in the area of cardiovascular implantable electronic device therapy is remote patient monitoring (RPM). RPM systems can interrogate the device automatically and send the data from the patients' home to the physician, thereby reducing in-clinic follow-ups.

The purpose of this study is to evaluate the effect of RPM + in-clinic follow-up versus in-clinic follow-up only on patient-reported health status and device-acceptance after implantation with an implantable cardioverter defibrillator (ICD) or cardiac resynchronization defibrillator (CRT-D).

Secondary objectives are (1) to identify subgroups of patients who prefer RPM over in-clinic visits or vice versa due to specific clinical and psychological factors and (2) To investigate the cost-effectiveness of RPM + in-clinic follow-up compared to in-clinic follow-up only.

ELIGIBILITY:
Inclusion Criteria:

* first time ICD/CRT-D implanted at one of the participating centers
* left ventricular ejection fraction <35%
* NYHA functional class II or III symptoms
* ICD/CRT-D device compatible with the LATITUDE(r) RPM system from Boston Scientific

Exclusion Criteria:

* On the waiting list for heart transplantation
* History of psychiatric illness others than affective/anxiety disorders
* Cognitive impairments
* Insufficient knowledge of the language to fill in the questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-04-13 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Patient-reported health status | 24 months
  23-item Kansas City Cardiomyopathy Questionnaire (KCCQ)
Patient-reported device acceptance | 24 months
  12-item Florida Patient Acceptance Scale (FPAS)

SECONDARY OUTCOMES:
Patient-reported satisfaction with care | 24 months
  * Visual Analogue Scale ranging from 0-100 (with higher score representing more satisfaction with care)
  * 26-item self-made questionnaire to assess satisfaction with RPM
Cost-effectiveness | 24 months
  Data regarding health care utilization is gathered from hospitals and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Meine, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] de Graaf G, Timmermans I, Meine M, Alings M, Pedersen SS, Mabo P, Zitron E, Redekop K, Versteeg H. Economic evaluation of remote monitoring of patients with an implantable cardiac defibrillator (REMOTE-CIED study). J Telemed Telecare. 2024 Aug;30(7):1173-1185. doi: 10.1177/1357633X221129176. Epub 2022 Oct 17. PMID 36245363
- [Derived] Chiu CSL, Timmermans I, Versteeg H, Zitron E, Mabo P, Pedersen SS, Meine M; REMOTE-CIED Trial Investigators. Effect of remote monitoring on clinical outcomes in European heart failure patients with an implantable cardioverter-defibrillator: secondary results of the REMOTE-CIED randomized trial. Europace. 2022 Feb 2;24(2):256-267. doi: 10.1093/europace/euab221. PMID 34410384
- [Derived] Versteeg H, Timmermans I, Widdershoven J, Kimman GJ, Prevot S, Rauwolf T, Scholten MF, Zitron E, Mabo P, Denollet J, Pedersen SS, Meine M. Effect of remote monitoring on patient-reported outcomes in European heart failure patients with an implantable cardioverter-defibrillator: primary results of the REMOTE-CIED randomized trial. Europace. 2019 Sep 1;21(9):1360-1368. doi: 10.1093/europace/euz140. PMID 31168604
- [Derived] Timmermans I, Meine M, Szendey I, Aring J, Romero Roldan J, van Erven L, Kahlert P, Zitron E, Mabo P, Denollet J, Versteeg H. Remote monitoring of implantable cardioverter defibrillators: Patient experiences and preferences for follow-up. Pacing Clin Electrophysiol. 2019 Feb;42(2):120-129. doi: 10.1111/pace.13574. Epub 2019 Jan 2. PMID 30536931
- [Derived] Timmermans I, Versteeg H, Meine M, Pedersen SS, Denollet J. Illness perceptions in patients with heart failure and an implantable cardioverter defibrillator: Dimensional structure, validity, and correlates of the brief illness perception questionnaire in Dutch, French and German patients. J Psychosom Res. 2017 Jun;97:1-8. doi: 10.1016/j.jpsychores.2017.03.014. Epub 2017 Mar 23. PMID 28606488